CLINICAL TRIAL: NCT06889857
Title: Safety and Efficacy of Intravenous Administration of SHED-CM for ALS
Acronym: SCA202401
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hitonowa Medical (Other)
Collaborators: U-Factor Co.,Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHED-CM-ALS-202401
Record Dates: First submitted 2024-07-18; First posted 2025-03-21 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS - Amyotrophic Lateral Sclerosis; Stem Cells; Conditioned Medium; Therapy; Safety; Regenerative Medicine
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: A group of ALS patients receiving the study drug
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Receiving the study drug (Experimental): The study drug will be administered intravenously at 120 ml once a week for 12 week.
  Interventions: Biological: The study drug is SHED-CM manufactured by U-Factor

INTERVENTIONS:
Biological: The study drug is SHED-CM manufactured by U-Factor — This study will involve informed consent, a 12-week observation period, a 12-week study drug administration period, and a 4-week follow-up period.

SUMMARY:
This study evaluates the safety and efficacy of Stem Cell from Human Exfoliated Deciduous teeth Conditioned Media (SHED-CM) in patients with Amyotrophic Lateral Sclerosis (ALS), using the Japanese version of the revised ALS Functional Rating Scale (ALSFRS-R) as an indicator.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the safety and efficacy of Stem Cell from Human Exfoliated Deciduous teeth Conditioned Media in patients with Amyotrophic Lateral Sclerosis (ALS), Particular focus will be placed on improving neurological function, slowing the rate of symptom progression, and improving the patient's quality of life.

What are the advantages of this therapy over standard therapy? and for which patients it is most effective ?

ELIGIBILITY:
Inclusion Criteria:

Patients who meet the following inclusion criteria (1) to (6) at the time of Informed consent

1. Patients who have provided written informed consent to participate in the study.
2. Patients who are at least 20 years of age at the time of obtaining informed consent.
3. Patients diagnosed with isolated or familial ALS and diagnosed as definite, the probable, or the probable laboratory-supported by updated Awaji criteria.
4. Patients with severity 1 or 2 on ALS severity criteria.
5. Outpatients.
6. Patients residing in Japan who can communicate in Japanese.

Exclusion Criteria:

Patients who do not meet any of the exclusion criteria (1) to (15) at the time of Informed consent

1. Patients with a tracheostomy
2. Patients with a history of non-invasive respiratory support
3. Patients with a percent FVC of 60 or less
4. Patients with chronic obstructive pulmonary disease (COPD)
5. Patients newly treated with edaravone or riluzole (oral) within 4 weeks prior to Informed consent
6. Patients receiving HAL medical leg type treatment
7. Patients receiving intravenous edaravone
8. Patients with cognitive impairment
9. Pregnant women or patients who may be pregnant
10. Patients with serious respiratory, cardiovascular, hepatic, or renal disease
11. Patients with malignant tumors
12. Patients with uncontrolled infection
13. Patients who have participated in other clinical trials within 12 weeks prior to obtaining consent
14. Patients with a history of drug allergy or severe allergic disease (e.g., anaphylactic shock) or concomitant history
15. Patients who are deemed inappropriate to participate in the study by the principal investigator or research coordinator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
All Adverse Events | Immediately after each administration and up to 4 weeks post-treatment
  This measure will check the total number of adverse events (AEs) reported during the study, categorized by CTCAE Ver 5.0 .
Number of Clinically Significant Changes in Laboratory Test Results | Baseline, Week 4, Week 8, Week 12, and at follow-up (Week 16).
  This measure will track the number of events where clinically significant abnormalities are detected in laboratory test parameters, including blood count, biochemistry, and coagulation function tests. Changes from baseline to follow-up are evaluated based on predefined clinical thresholds.
Number of Clinically Significant Changes in Vital Signs | Baseline, Week 4, Week 8, Week 12, and at follow-up (Week 16).
  This measure will evaluate the number of events where clinically significant changes in vital signs occur. Parameters include systolic blood pressure, diastolic blood pressure, pulse rate, body temperature, and SpO2. Each event will be assessed at two time points: immediately after treatment and after follow-up session, comparing values to baseline.
Safety assessment during the study period: Adverse events - Self- and other findings | Immediately after each administration and up to 4 weeks post-treatment
  Medical examination, subjective findings, Other findings

SECONDARY OUTCOMES:
Efficacy assessment: ALSFRS-R | Change from baseline ALSFRS-R at follow-up session
  The revised ALS Functional Rating Scale in ALS Patients. This scale is scored from 0 to 48, the higher the score the better.
Efficacy assessment: %FVC | Change from baseline %FVC at follow-up session
  % forced vital capacity in ALS Patients
Efficacy assessment: grip strength | Change from baseline grip strength at follow-up session
  grip strength in ALS Patients

CONTACTS AND LOCATIONS:
Locations (1):
- Hitonowa Medical, Chiyoda City, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oki R, Izumi Y, Fujita K, Miyamoto R, Nodera H, Sato Y, Sakaguchi S, Nokihara H, Kanai K, Tsunemi T, Hattori N, Hatanaka Y, Sonoo M, Atsuta N, Sobue G, Shimizu T, Shibuya K, Ikeda K, Kano O, Nishinaka K, Kojima Y, Oda M, Komai K, Kikuchi H, Kohara N, Urushitani M, Nakayama Y, Ito H, Nagai M, Nishiyama K, Kuzume D, Shimohama S, Shimohata T, Abe K, Ishihara T, Onodera O, Isose S, Araki N, Morita M, Noda K, Toda T, Maruyama H, Furuya H, Teramukai S, Kagimura T, Noma K, Yanagawa H, Kuwabara S, Kaji R; Japan Early-Stage Trial of Ultrahigh-Dose Methylcobalamin for ALS (JETALS) Collaborators. Efficacy and Safety of Ultrahigh-Dose Methylcobalamin in Early-Stage Amyotrophic Lateral Sclerosis: A Randomized Clinical Trial. JAMA Neurol. 2022 Jun 1;79(6):575-583. doi: 10.1001/jamaneurol.2022.0901. PMID 35532908
- See also: We referenced this paper because of the Phase III trial in ALS. — https://pubmed.ncbi.nlm.nih.gov/35532908/